CLINICAL TRIAL: NCT00541658
Title: A Non-inferiority Comparison of 35 mg Delayed-release Risedronate, Given Once-weekly Either Before or After Breakfast, & 5 mg Immediate-release Risedronate, Given Once-daily Before Breakfast, in the Treatment of Postmenopausal Osteoporosis.
Brief Title: A Study of a 35 mg Delayed Release Formulation of Risedronate for Osteoporosis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Warner Chilcott (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2007008
Record Dates: First submitted 2007-10-05; First posted 2007-10-10 (Estimated); Results first posted 2011-06-21 (Estimated); Last update posted 2013-04-22 (Estimated); Status verified 2013-04

CONDITIONS: Postmenopausal Osteoporosis
MeSH Terms: conditions — Osteoporosis, Postmenopausal | interventions — Risedronic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- 5 mg Before Breakfast (Active Comparator): 5 mg / Immediate-release Risedronate (At Least 30 Minutes Before Breakfast)
  Interventions: Drug: risedronate
- 35 mg After Breakfast (Experimental): 35 mg / Delayed-release Risedronate (Immediately Following Breakfast)
  Interventions: Drug: risedronate
- 35 mg Before Breakfast (Experimental): 35 mg / Delayed-release Risedronate (At Least 30 Minutes Before Breakfast)
  Interventions: Drug: risedronate

INTERVENTIONS:
Drug: risedronate — 5 mg Immediate-release Risedronate Administered At Least 30 Minutes Before Breakfast Daily
  Other Names: IRBB
  Arms: 5 mg Before Breakfast
Drug: risedronate — 35 mg Delayed-release Risedronate Administered Immediately Following Breakfast Weekly
  Other Names: DRFB
  Arms: 35 mg After Breakfast
Drug: risedronate — 35 mg Delayed-release Risedronate Administered At Least 30 Minutes Before Breakfast Weekly
  Other Names: DRBB
  Arms: 35 mg Before Breakfast

SUMMARY:
The purpose of this trial is to study the efficacy of a 35 mg delayed release weekly dosing regimen as compared to the standard daily dosing regimen of risedronate 5 mg daily.

DETAILED DESCRIPTION:
The comparator arms of this risedronate study are 35 mg delayed release given weekly and 5 mg immediate release given daily.

ELIGIBILITY:
Inclusion Criteria:

* Female: 50 years of age or older
* >5 years since last menses natural or surgical
* have lumbar spine or total hip BMD more that 2.5 SD below the young adult mean, or have lumbar spine or total hip BMD more than 2.0 SD below the young adult female mean value and also have at least one prevalent vertebral body fracture

Exclusion Criteria:

* history of uncontrolled hyperparathyroidism, hyperthyroidism, osteomalacia
* BMI >32 kg/m
* use of medications within 3 months of starting study drug that impact bone metabolism such as glucocorticoids, estrogens, calcitonin, calcitriol, other bisphosphonates and parathyroid hormone
* hypocalcemia or hypercalcemia of any cause
* markedly abnormal clinical laboratory measurements that are assessed as clinically significant by the investigator

Min Age: 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 923 (Actual)
Dates: Start 2007-10; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ana Balske, MD, PhD, Study Director — Procter and Gamble
Locations (45):
- United States (20):
  - Research Site, Birmingham, Alabama
  - Research Site, Oakland, California
  - Research Site, San Diego, California
  - Research Facility, Walnut Creek, California
  - Research Site, Walnut Creek, California
  - Research Site, Lakewood, Colorado
  - Research Site, Leesburg, Florida
  - Research Site, Melbourne, Florida
  - Research Site, South Miami, Florida
  - Research Site, Gainesville, Georgia
  - Research Site, Champaign, Illinois
  - Research Site, Chicago, Illinois
  - Research Site, Bethesda, Maryland
  - Research Site, Brockton, Massachusetts
  - Research Site, Omaha, Nebraska
  - Research Site, Las Vegas, Nevada
  - Research Site, Greenville, North Carolina
  - Research Site, Portland, Oregon
  - Research Site, Seattle, Washington
  - Research Site, Madison, Wisconsin
- Research Site, Buenos Aires, Argentina
- Belgium (3):
  - Research Facility, Diepenbeek
  - Research Site, Ghent
  - Research Site, Leuven
- Canada (7):
  - Research Site, Hamilton, Ontario
  - Research Site, Kitchener, Ontario
  - Research Site, Newmarket, Ontario
  - Research Site, Montreal, Quebec
  - Research Site, Québec, Quebec
  - Research Site, Saint-Eustache, Quebec
  - Research Site, Saskatoon, Saskatchewan
- Estonia (3):
  - Research Site, Pärnu
  - Research Site, Tallinn
  - Research Site, Tartu
- France (4):
  - Research Site, Amiens
  - Research Site, Lyon
  - Research Site, Orléans
  - Research Site, Vandœuvre-lès-Nancy
- Hungary (5):
  - Research Site, Balatonfüred
  - Research Site, Debrecen
  - Research Site, Eger
  - Research Site, Győr
  - Research Site, Koranyi Sandor
- Poland (2):
  - Research Site, Bialystok
  - Research Site, Warsaw

REFERENCES:
- [Derived] McClung MR, Miller PD, Brown JP, Zanchetta J, Bolognese MA, Benhamou CL, Balske A, Burgio DE, Sarley J, McCullough LK, Recker RR. Efficacy and safety of a novel delayed-release risedronate 35 mg once-a-week tablet. Osteoporos Int. 2012 Jan;23(1):267-76. doi: 10.1007/s00198-011-1791-y. Epub 2011 Sep 27. PMID 21947137

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 923 women with PMO at 43 sites in 8 countries across North America, South America, and the European Union. Patients were randomized within a site to 1 of 3 treatment groups (35 mg delayed-release Risedronate, given once-weekly before/after breakfast, and 5 mg immediate-release Risedronate, administered once-daily before breakfast) in a 1:1:1 ratio.
Groups:
- 5 mg Before Breakfast: 5 mg risedronate immediate-release daily tablet administered at least 30 minutes before breakfast (IRBB)
- 35 mg After Breakfast: 35 mg risedronate delayed-release immediately following breakfast (DRFB), administered once-a-week
- 35 mg Before Breakfast: 35 mg risedronate delayed-release administered at least 30 minutes before breakfast (DRBB), once-a-week
Period: Overall Study
Arm/Group | 5 mg Before Breakfast | 35 mg After Breakfast | 35 mg Before Breakfast
Started | 308 | 307 | 308
ITT Population | 307 | 307 | 308
Completed | 248 | 234 | 240
Not Completed | 60 | 73 | 68
Not completed — Adverse Event | 28 | 37 | 25
Not completed — Physician Decision | 0 | 0 | 4
Not completed — Lost to Follow-up | 3 | 3 | 6
Not completed — Protocol Violation | 0 | 1 | 1
Not completed — Withdrawal by Subject | 28 | 32 | 32
Not completed — Took No Study Drug | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 5 mg Before Breakfast | 35 mg After Breakfast | 35 mg Before Breakfast | Total
Number analyzed (Participants) | 308 | 307 | 308 | 923
Age Continuous [Mean (Standard Deviation); unit: years] — ITT Population
  years | 65.3 (7.4) | 65.8 (7.4) | 66.0 (7.5) | 65.7 (7.4)
Age, Customized [Number; unit: participants] — ITT Population
  participants
    < 65 years | 141 | 127 | 133 | 401
    Between 65 and < 75 years | 128 | 141 | 133 | 402
    > = 75 years | 38 | 39 | 42 | 119
Gender [Number; unit: participants] — ITT Population
  participants
    Female | 307 | 307 | 308 | 922
    Male | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Argentina | 88 | 85 | 84 | 257
  Belgium | 4 | 5 | 3 | 12
  Canada | 7 | 7 | 9 | 23
  Estonia | 53 | 53 | 52 | 158
  France | 19 | 23 | 18 | 60
  Hungary | 35 | 34 | 33 | 102
  Poland | 56 | 57 | 58 | 171
  United States | 46 | 43 | 51 | 140

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline Lumbar Spine Bone Mineral Density (BMD) at Week 52 / Endpoint, ITT Population
Time Frame: 52 weeks / Endpoint
Population: Intention-to-Treat (ITT) Population. Last Observation Carried Forward (LOCF) at Week 52.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent Change
Arm/Group | 5 mg Before Breakfast | 35 mg After Breakfast | 35 mg Before Breakfast
Number analyzed (Participants) | 270 | 261 | 271
Percent Change | 3.069 [2.664 to 3.474] | 3.302 [2.890 to 3.715] | 3.365 [2.961 to 3.769]
Statistical Analysis 1: Comparison: 5 mg Before Breakfast vs 35 mg After Breakfast; Test type: Non-Inferiority or Equivalence — To establish the non-inferiority at one-sided α of 2.5% with 90% power, 651 patients (217 per treatment group) was required to complete at least 52 weeks of the study. Adjusting for 20% dropouts, 272 patients per group were required for randomization. This calculation was based on a non-inferiority margin of 1.5%, a true mean difference (μIR - μDR) of 0.25%, and a common standard deviation of the percent change from baseline in lumbar spine BMD at Week 52 of 4.0%; ANOVA; Fixed effects for treatment, pooled center and anticoagulant use; Least Squares Mean Difference = -0.233, 95% CI 2-sided [-0.812 to 0.345] — LS Mean Difference is 5 mg daily minus weekly treatment
Statistical Analysis 2: Comparison: 5 mg Before Breakfast vs 35 mg Before Breakfast; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; ANOVA; Fixed effects for treatment, pooled center and anticoagulant use; Least Squares Mean Difference = -0.296, 95% CI 2-sided [-0.869 to 0.277] — LS Mean Difference is 5 mg daily minus weekly treatment

2. Secondary Outcome: Percent Change From Baseline Lumbar Spine BMD for Combined 35 mg Delayed-Release Weekly Treatment Group, Week 52 / Endpoint, ITT Population
Time Frame: Week 52 / Endpoint
Population: 35 mg group combined delayed-relase following breakfast (DRFB) group with delayed-relase before breakfast (DRBB) group and compared with 5 mg immediate-release before breakfast (IRBB) group. ITT Population. Last Observation Carried Forward at Week 52.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent Change
Groups:
- 5 mg IRBB: 5 mg immediate-release risedronate tablet daily, at least 30 minutes before breakfast for two years
- 35 mg DRFB + DRBB: Combined two arms - 35 mg delayed-release following breakfast (DRFB) with 35 mg delayed-relase before breakfast (DRBB)
Arm/Group | 5 mg IRBB | 35 mg DRFB + DRBB
Number analyzed (Participants) | 270 | 532
Percent Change | 3.069 [2.664 to 3.474] | 3.334 [3.046 to 3.622]
Statistical Analysis 1: Comparison: 5 mg IRBB vs 35 mg DRFB + DRBB; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.2955, ANOVA; Fixed effects for treatment, pooled center and anticoagulant used; Least Squares Mean Difference = -0.265, 95% CI 2-sided [-0.763 to 0.232] — LS Mean Difference is 5 mg daily minus weekly treatment

3. Secondary Outcome: Percent Change From Baseline Lumbar Spine BMD, Week 26, ITT Population
Time Frame: Week 26
Population: ITT Population
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent Change
Arm/Group | 5 mg Before Breakfast | 35 mg After Breakfast | 35 mg Before Breakfast
Number analyzed (Participants) | 269 | 261 | 269
Percent Change | 2.685 [2.305 to 3.066] | 2.816 [2.429 to 3.203] | 2.529 [2.148 to 2.910]
Statistical Analysis 1: Comparison: 5 mg Before Breakfast vs 35 mg After Breakfast; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; ANOVA; Fixed effects for treatment, pooled center and anticoagulant use; Least Squares Mean Difference = -0.131, 95% CI 2-sided [-0.674 to 0.412] — LS Mean Difference is 5 mg daily minus weekly treatment
Statistical Analysis 2: Comparison: 5 mg Before Breakfast vs 35 mg Before Breakfast; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; ANOVA; Fixed effects for treatment, pooled center and anticoagulant use; Least Squares Mean Difference = 0.156, 95% CI 2-sided [-0.382 to 0.695] — LS Mean Difference is 5 mg daily minus weekly treatment

4. Secondary Outcome: Percent Change From Baseline Lumbar Spine BMD, Week 52, ITT Population
Time Frame: Week 52
Population: ITT Population
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent Change
Arm/Group | 5 mg Before Breakfast | 35 mg After Breakfast | 35 mg Before Breakfast
Number analyzed (Participants) | 258 | 257 | 258
Percent Change | 3.035 [2.627 to 3.443] | 3.293 [2.883 to 3.702] | 3.357 [2.949 to 3.766]
Statistical Analysis 1: Comparison: 5 mg Before Breakfast vs 35 mg After Breakfast; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; ANOVA; Fixed effects for treatment, pooled center and anticoagulant use; Least Squares Mean Difference = -0.258, 95% CI 2-sided [-0.836 to 0.321] — LS Mean Difference is 5 mg daily minus weekly treatment
Statistical Analysis 2: Comparison: 5 mg Before Breakfast vs 35 mg Before Breakfast; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; ANOVA; Fixed effects for treatment, pooled center and anticoagulant use; Least Squares Mean Difference = -0.322, 95% CI 2-sided [-0.900 to 0.256] — LS Mean Difference is 5 mg daily minus weekly treatment

5. Secondary Outcome: Percent Change From Baseline Lumbar Spine BMD at Week 104, ITT Population
Time Frame: Week 104
Population: ITT Population
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent Change
Arm/Group | 5 mg Before Breakfast | 35 mg After Breakfast | 35 mg Before Breakfast
Number analyzed (Participants) | 242 | 232 | 235
Percent Change | 4.352 [3.829 to 4.874] | 5.506 [4.971 to 6.040] | 5.396 [4.865 to 5.926]
Statistical Analysis 1: Comparison: 5 mg Before Breakfast vs 35 mg After Breakfast; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; ANOVA; Fixed effects for treatment, pooled center and anticoagulant use; LS Mean Difference = -1.154, 95% CI 2-sided [-1.903 to -0.405] — LS Mean Difference is 5 mg daily minus weekly treatment
Statistical Analysis 2: Comparison: 5 mg Before Breakfast vs 35 mg Before Breakfast; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; ANOVA; Fixed effects for treatment, pooled center and anticoagulant use; LS Mean Difference = -1.044, 95% CI 2-sided [-1.789 to -0.299] — LS Mean Difference is 5 mg daily minus weekly treatment

6. Secondary Outcome: Percent Change From Baseline Lumbar Spine BMD at Week 104 / Endpoint, ITT Population
Time Frame: Week 104 / Endpoint
Population: ITT Population. Last Observation Carried Forward at Week 104.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent Change
Arm/Group | 5 mg Before Breakfast | 35 mg After Breakfast | 35 mg Before Breakfast
Number analyzed (Participants) | 274 | 265 | 273
Percent Change | 4.147 [3.653 to 4.640] | 5.205 [4.703 to 5.707] | 5.068 [4.574 to 5.562]
Statistical Analysis 1: Comparison: 5 mg Before Breakfast vs 35 mg After Breakfast; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; ANOVA; Fixed effects for treatment, pooled center and anticoagulant use; LS Mean Difference = -1.059, 95% CI 2-sided [-1.762 to -0.355] — LS Mean Difference is 5 mg daily minus weekly treatment
Statistical Analysis 2: Comparison: 5 mg Before Breakfast vs 35 mg Before Breakfast; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; ANOVA; Fixed effects for treatment, pooled center and anticoagulant use; LS Mean Difference = -0.922, 95% CI 2-sided [-1.620 to -0.223] — LS Mean Difference is 5 mg daily minus weekly treatment

7. Secondary Outcome: Percent Responders to Treatment (>0% Change From Baseline in Lumbar Spine BMD), Week 52, ITT Population
Description: Responder = a patient showing a positive change (>0 g/cm2) in lumbar spine BMD from baseline to the timepoint.
Time Frame: Week 52
Population: ITT Population.
Measure: Number; unit: Percentage of Participants
Arm/Group | 5 mg Before Breakfast | 35 mg After Breakfast | 35 mg Before Breakfast
Number analyzed (Participants) | 258 | 257 | 258
Percentage of Participants | 81 | 87.5 | 86.4
Statistical Analysis 1: Comparison: 5 mg Before Breakfast vs 35 mg After Breakfast; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.0524, Fisher Exact; Relative Risk = 1.08, 95% CI 2-sided [1.00 to 1.16]
Statistical Analysis 2: Comparison: 5 mg Before Breakfast vs 35 mg Before Breakfast; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.1207, Fisher Exact; Relative Risk = 1.07, 95% CI 2-sided [0.99 to 1.15]

8. Secondary Outcome: Percent Responders to Treatment (>0% Change From Baseline in Lumbar Spine BMD) at Week 52 / Endpoint, ITT Population
Description: Responder = a patient showing a positive change (>0 g/cm2) in lumbar spine BMD from baseline to the timepoint.
Time Frame: Week 52 / Endpoint
Population: ITT Population. Last Observation Carried Forward at Week 52.
Measure: Number; unit: Percentage of Participants
Arm/Group | 5 mg Before Breakfast | 35 mg After Breakfast | 35 mg Before Breakfast
Number analyzed (Participants) | 270 | 261 | 271
Percentage of Participants | 81.5 | 87.4 | 86.0
Statistical Analysis 1: Comparison: 5 mg Before Breakfast vs 35 mg After Breakfast; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.0729, Fisher Exact; Relative Risk = 1.07, 95% CI 2-sided [1.00 to 1.15]
Statistical Analysis 2: Comparison: 5 mg Before Breakfast vs 35 mg Before Breakfast; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.1639, Fisher Exact; Relative Risk = 1.06, 95% CI 2-sided [0.98 to 1.14]

9. Secondary Outcome: Percent Responders to Treatment (>0% Change From Baseline in Lumbar Spine BMD) at Week 104, ITT Population
Description: Responder = a patient showing a positive change (>0 g/cm2) in lumbar spine BMD from baseline to the timepoint.
Time Frame: Week 52
Population: ITT Population
Measure: Number; unit: Percentage of Participants
Arm/Group | 5 mg Before Breakfast | 35 mg After Breakfast | 35 mg Before Breakfast
Number analyzed (Participants) | 242 | 232 | 235
Percentage of Participants | 82.6 | 89.2 | 92.3
Statistical Analysis 1: Comparison: 5 mg Before Breakfast vs 35 mg After Breakfast; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.0476, Fisher Exact; Relative Risk = 1.08, 95% CI 2-sided [1.00 to 1.16]
Statistical Analysis 2: Comparison: 5 mg Before Breakfast vs 35 mg Before Breakfast; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.0014, ANOVA; Relative Risk = 1.12, 95% CI 2-sided [1.04 to 1.20]

10. Secondary Outcome: Percent Responders to Treatment (>0% Change From Baseline in Lumbar Spine BMD) at Week 104 / Endpoint, ITT Population
Description: Responder = a patient showing a positive change (>0 g/cm2) in lumbar spine BMD from baseline to the timepoint.
Time Frame: Week 52 / Endpoint
Population: ITT Population. Last Observation Carried Forward at Week 104.
Measure: Number; unit: Percentage of Participants
Arm/Group | 5 mg Before Breakfast | 35 mg After Breakfast | 35 mg Before Breakfast
Number analyzed (Participants) | 274 | 265 | 273
Percentage of Participants | 81.8 | 87.9 | 90.1
Statistical Analysis 1: Comparison: 5 mg Before Breakfast vs 35 mg After Breakfast; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.0547, ANOVA; Relative Risk = 1.08, 95% CI 2-sided [1.00 to 1.16]
Statistical Analysis 2: Comparison: 5 mg Before Breakfast vs 35 mg Before Breakfast; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.0066, ANOVA; Relative Risk = 1.10, 95% CI 2-sided [1.03 to 1.18]

11. Secondary Outcome: Percent Change From Baseline in Total Proximal Femur BMD, Week 26, ITT Population
Time Frame: Week 26
Population: ITT Population.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent Change
Arm/Group | 5 mg Before Breakfast | 35 mg After Breakfast | 35 mg Before Breakfast
Number analyzed (Participants) | 273 | 267 | 275
Percent Change | 1.613 [1.354 to 1.872] | 1.748 [1.486 to 2.010] | 1.685 [1.426 to 1.943]
Statistical Analysis 1: Comparison: 5 mg Before Breakfast vs 35 mg After Breakfast; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; ANOVA; Fixed effect for treatment, pooled center and anticoagulant use; Least Squares Mean Difference = -0.135, 95% CI 2-sided [-0.504 to 0.234] — LS Mean Difference is 5 mg daily minus weekly treatment
Statistical Analysis 2: Comparison: 5 mg Before Breakfast vs 35 mg Before Breakfast; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; ANOVA; Fixed effect for treatment, pooled center and anticoagulant use; Least Squares Mean Difference = -0.072, 95% CI 2-sided [-0.437 to 0.294] — LS Mean Difference is 5 mg daily minus weekly treatment

12. Secondary Outcome: Percent Change From Baseline in Total Proximal Femur BMD, Week 52, ITT Population
Time Frame: Week 52
Population: ITT Population.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent
Arm/Group | 5 mg Before Breakfast | 35 mg After Breakfast | 35 mg Before Breakfast
Number analyzed (Participants) | 258 | 256 | 258
Percent | 1.809 [1.524 to 2.093] | 2.130 [1.845 to 2.415] | 2.099 [1.815 to 2.383]
Statistical Analysis 1: Comparison: 5 mg Before Breakfast vs 35 mg After Breakfast; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; ANOVA; Fixed effects for treatment, pooled center and anticoagulant use; Least Squares Mean Difference = -0.321, 95% CI 2-sided [-0.724 to 0.082] — LS Mean Difference is 5 mg daily minus weekly treatment
Statistical Analysis 2: Comparison: 5 mg Before Breakfast vs 35 mg Before Breakfast; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; ANOVA; Fixed effects for treatment, pooled center and anticoagulant use; Least Squares Mean Difference = -0.290, 95% CI 2-sided [-0.692 to 0.112] — LS Mean Difference is 5 mg daily minus weekly treatment

13. Secondary Outcome: Percent Change From Baseline Total Proximal Femur BMD, Week 52 / Endpoint, ITT Population
Time Frame: Week 52 / Endpoint
Population: ITT Population. Last Observation Carried Forward at Week 52.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent Change
Arm/Group | 5 mg Before Breakfast | 35 mg After Breakfast | 35 mg Before Breakfast
Number analyzed (Participants) | 279 | 274 | 280
Percent Change | 1.785 [1.508 to 2.062] | 2.073 [1.793 to 2.352] | 2.075 [1.799 to 2.352]
Statistical Analysis 1: Comparison: 5 mg Before Breakfast vs 35 mg After Breakfast; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; ANOVA; Fixed effect for treatment, pooled center and anticoagulant use; Least Squares Mean Difference = -0.288, 95% CI 2-sided [-0.682 to 0.106] — LS Mean Difference is 5 mg daily minus weekly treatment
Statistical Analysis 2: Comparison: 5 mg Before Breakfast vs 35 mg Before Breakfast; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; ANOVA; Fixed effects for treatment, pooled center and anticoagulant use; Least Squares Mean Difference = -0.290, 95% CI 2-sided [-0.681 to 0.101] — LS Mean Difference is 5 mg daily minus weekly treatment

14. Secondary Outcome: Percent Change From Baseline Total Proximal Femur BMD, Week 104, ITT Population
Time Frame: Week 104
Population: ITT Population
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent Change
Arm/Group | 5 mg Before Breakfast | 35 mg After Breakfast | 35 mg Before Breakfast
Number analyzed (Participants) | 244 | 231 | 239
Percent Change | 2.177 [1.805 to 2.549] | 2.821 [2.438 to 3.204] | 2.764 [2.389 to 3.140]
Statistical Analysis 1: Comparison: 5 mg Before Breakfast vs 35 mg After Breakfast; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; ANOVA; LS Mean Difference = -0.644, 95% CI 2-sided [-1.179 to -0.110]
Statistical Analysis 2: Comparison: 5 mg Before Breakfast vs 35 mg Before Breakfast; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; ANOVA; LS Mean Difference = -0.587, 95% CI 2-sided [-1.116 to -0.059]

15. Secondary Outcome: Percent Change From Baseline Total Proximal Femur BMD, Week 104 / Endpoint, ITT Population
Time Frame: Week 104 / Endpoint
Population: ITT Population. Last Observation Carried Forward at Week 104.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent Change
Arm/Group | 5 mg Before Breakfast | 35 mg After Breakfast | 35 mg Before Breakfast
Number analyzed (Participants) | 279 | 274 | 280
Percent Change | 2.028 [1.671 to 2.386] | 2.551 [2.190 to 2.912] | 2.496 [2.139 to 2.853]
Statistical Analysis 1: Comparison: 5 mg Before Breakfast vs 35 mg After Breakfast; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; ANOVA; LS Mean Difference = -0.522, 95% CI 2-sided [-1.030 to -0.014]
Statistical Analysis 2: Comparison: 5 mg Before Breakfast vs 35 mg Before Breakfast; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; ANOVA; LS Mean Difference = -0.468, 95% CI 2-sided [-0.973 to 0.037]

16. Secondary Outcome: Percent Change From Baseline in Femoral Neck BMD, Week 26, ITT Population
Time Frame: Week 26
Population: ITT Population
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent Change
Arm/Group | 5 mg Before Breakfast | 35 mg After Breakfast | 35 mg Before Breakfast
Number analyzed (Participants) | 273 | 267 | 275
Percent Change | 1.120 [0.792 to 1.447] | 1.385 [1.053 to 1.716] | 1.246 [0.920 to 1.572]
Statistical Analysis 1: Comparison: 5 mg Before Breakfast vs 35 mg After Breakfast; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; ANOVA; Fixed effects for treatment, pooled centers and anticoagulant use; Least Squares Mean Difference = -0.265, 95% CI 2-sided [-0.731 to 0.201] — LS Mean Difference is 5 mg daily minus weekly treatment
Statistical Analysis 2: Comparison: 5 mg Before Breakfast vs 35 mg Before Breakfast; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; ANOVA; Fixed effects for treatment, pooled center and anticoagulant use; Least Squares Mean Difference = -0.126, 95% CI 2-sided [-0.588 to 0.336] — LS Mean Difference is 5 mg daily minus weekly treatment

17. Secondary Outcome: Percent Change From Baseline in Femoral Neck BMD, Week 52, ITT Population
Time Frame: Week 52
Population: ITT Population
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent Change
Arm/Group | 5 mg Before Breakfast | 35 mg After Breakfast | 35 mg Before Breakfast
Number analyzed (Participants) | 258 | 256 | 258
Percent Change | 1.155 [0.814 to 1.496] | 1.482 [1.140 to 1.825] | 1.717 [1.376 to 2.058]
Statistical Analysis 1: Comparison: 5 mg Before Breakfast vs 35 mg After Breakfast; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; ANOVA; Fixed effects for treatment, pooled centers and anticoagulant use; Least Squares Mean Difference = -0.328, 95% CI 2-sided [-0.811 to 0.156] — LS Mean Difference is 5 mg daily minus weekly treatment
Statistical Analysis 2: Comparison: 5 mg Before Breakfast vs 35 mg Before Breakfast; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; ANOVA; Fixed effects for treatment, pooled center, anticoagulant use; Least Squares Mean Difference = -0.563, 95% CI 2-sided [-1.045 to -0.080] — LS Mean Difference is 5 mg daily minus weekly treatment

18. Secondary Outcome: Percent Change From Baseline in Femoral Neck BMD, Week 52 / Endpoint, ITT Population
Time Frame: Week 52 / Endpoint
Population: ITT Population. LOCF at Week 52.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent Change
Arm/Group | 5 mg Before Breakfast | 35 mg After Breakfast | 35 mg Before Breakfast
Number analyzed (Participants) | 279 | 274 | 280
Percent Change | 1.180 [0.853 to 1.507] | 1.507 [1.177 to 1.838] | 1.717 [1.390 to 2.044]
Statistical Analysis 1: Comparison: 5 mg Before Breakfast vs 35 mg After Breakfast; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; ANOVA; Fixed effects for treatment, pooled center and anticoagulant use; Least Squares Mean Difference = -0.327, 95% CI 2-sided [-0.793 to 0.138] — LS Mean Difference is 5 mg daily minus weekly treatment
Statistical Analysis 2: Comparison: 5 mg Before Breakfast vs 35 mg Before Breakfast; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; ANOVA; Fixed effects for treatment, pooled center and anticoagulant use; Least Squares Mean Difference = -0.537, 95% CI 2-sided [-1.000 to -0.074] — LS Mean Difference is 5 mg daily minus weekly treatment

19. Secondary Outcome: Percent Change From Baseline in Femoral Neck BMD, Week 104, ITT Population
Time Frame: Week 104
Population: ITT Population
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent Change
Arm/Group | 5 mg Before Breakfast | 35 mg After Breakfast | 35 mg Before Breakfast
Number analyzed (Participants) | 244 | 231 | 239
Percent Change | 1.530 [1.105 to 1.955] | 2.108 [1.670 to 2.545] | 2.328 [1.899 to 2.758]
Statistical Analysis 1: Comparison: 5 mg Before Breakfast vs 35 mg After Breakfast; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; ANOVA; Fixed effects for treatment, pooled center and anticoagulant use; LS Mean Difference = -0.578, 95% CI 2-sided [-1.189 to 0.032] — LS Mean Difference is 5 mg daily minus weekly treatment
Statistical Analysis 2: Comparison: 5 mg Before Breakfast vs 35 mg Before Breakfast; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; ANOVA; Fixed effects for treatment, pooled center and anticoagulant use; LS Mean Difference = -0.799, 95% CI 2-sided [-1.403 to -0.194] — LS Mean Difference is 5 mg daily minus weekly treatment

20. Secondary Outcome: Percent Change From Baseline in Femoral Neck BMD, Week 104 / Endpoint, ITT Population
Time Frame: Week 104 / Endpoint
Population: ITT Population. LOCF at Week 104.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent Change
Arm/Group | 5 mg Before Breakfast | 35 mg After Breakfast | 35 mg Before Breakfast
Number analyzed (Participants) | 279 | 274 | 280
Percent Change | 1.431 [1.028 to 1.834] | 1.986 [1.579 to 2.393] | 2.047 [1.644 to 2.449]
Statistical Analysis 1: Comparison: 5 mg Before Breakfast vs 35 mg After Breakfast; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; ANOVA; Fixed effects for treatment, pooled center and anticoagulant use; LS Mean Difference = -0.555, 95% CI 2-sided [-1.128 to 0.018] — LS Mean Difference is 5 mg daily minus weekly treatment
Statistical Analysis 2: Comparison: 5 mg Before Breakfast vs 35 mg Before Breakfast; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; ANOVA; Fixed effect for treatment, pooled center and anticoagulant use; LS Mean Difference = -0.616, 95% CI 2-sided [-1.185 to -0.046] — LS Mean Difference is 5 mg daily minus weekly treatment

21. Secondary Outcome: Percent Change From Baseline Greater Trochanter BMD, Week 26, ITT Population
Time Frame: Week 26
Population: ITT Population.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent Change
Arm/Group | 5 mg Before Breakfast | 35 mg After Breakfast | 35 mg Before Breakfast
Number analyzed (Participants) | 273 | 267 | 275
Percent Change | 1.900 [1.470 to 2.329] | 2.148 [1.713 to 2.583] | 2.164 [1.736 to 2.592]
Statistical Analysis 1: Comparison: 5 mg Before Breakfast vs 35 mg After Breakfast; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; ANOVA; Fixed effects for treatment, pooled center and anticoagulant use; Least Squares Mean Difference = -0.249, 95% CI 2-sided [-0.860 to 0.363] — LS Mean Difference is 5 mg daily minus weekly treatment
Statistical Analysis 2: Comparison: 5 mg Before Breakfast vs 35 mg Before Breakfast; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; ANOVA; Fixed effect for treatment, pooled center and anticoagulant use; Least Squares Mean Difference = -0.265, 95% CI 2-sided [-0.871 to 0.342] — LS Mean Difference is 5 mg daily minus weekly treatment

22. Secondary Outcome: Percent Change From Baseline in Greater Trochanter BMD, Week 52, ITT Population
Time Frame: Week 52
Population: ITT Population.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent Change
Arm/Group | 5 mg Before Breakfast | 35 mg After Breakfast | 35 mg Before Breakfast
Number analyzed (Participants) | 258 | 256 | 258
Percent Change | 2.297 [1.854 to 2.740] | 2.854 [2.409 to 3.299] | 2.819 [2.376 to 3.262]
Statistical Analysis 1: Comparison: 5 mg Before Breakfast vs 35 mg After Breakfast; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; ANOVA; Fixed effects for treatment, pooled center and anticoagulant use; Least Squares Mean Difference = -0.557, 95% CI 2-sided [-1.185 to 0.071] — LS Mean Difference is 5 mg daily minus weekly treatment
Statistical Analysis 2: Comparison: 5 mg Before Breakfast vs 35 mg Before Breakfast; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; ANOVA; Least Squares Mean Difference = -0.522, 95% CI 2-sided [-1.149 to 0.105] — LS Mean Difference is 5 mg daily minus weekly treatment

23. Secondary Outcome: Percent Change From Baseline in Greater Trochanter BMD, Week 52 / Endpoint
Time Frame: Week 52 / Endpoint
Population: ITT Population. Last Observation Carried Forward at Week 52.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent Change
Arm/Group | 5 mg Before Breakfast | 35 mg After Breakfast | 35 mg Before Breakfast
Number analyzed (Participants) | 279 | 274 | 280
Percent Change | 2.186 [1.746 to 2.625] | 2.732 [2.288 to 3.175] | 2.764 [2.326 to 3.203]
Statistical Analysis 1: Comparison: 5 mg Before Breakfast vs 35 mg After Breakfast; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; ANOVA; Fixed effects for treatment, pooled center and anticoagulant use; Least Squares Mean Difference = -0.546, 95% CI 2-sided [-1.170 to 0.078] — LS Mean Difference is 5 mg daily minus weekly treatment
Statistical Analysis 2: Comparison: 5 mg Before Breakfast vs 35 mg Before Breakfast; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; ANOVA; Fixed effects for treatment, pooled center and anticoagulant use; Least Squares Mean Difference = -0.579, 95% CI 2-sided [-1.199 to 0.042] — LS Mean Difference is 5 mg daily minus weekly treatment

24. Secondary Outcome: Percent Change From Baseline in Greater Trochanter BMD, Week 104, ITT Population
Time Frame: Week 104
Population: ITT Population.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent Change
Arm/Group | 5 mg Before Breakfast | 35 mg After Breakfast | 35 mg Before Breakfast
Number analyzed (Participants) | 244 | 231 | 239
Percent Change | 3.056 [2.523 to 3.589] | 4.152 [3.603 to 4.700] | 4.246 [3.707 to 4.785]
Statistical Analysis 1: Comparison: 5 mg Before Breakfast vs 35 mg After Breakfast; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; ANOVA; Fixed effects for treatment, pooled center and anticoagulant use; LS Mean Difference = -1.095, 95% CI 2-sided [-1.861 to -0.329] — LS Mean Difference is 5 mg daily minus weekly treatment
Statistical Analysis 2: Comparison: 5 mg Before Breakfast vs 35 mg Before Breakfast; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; ANOVA; Fixed effects for treatment, pooled center and anticoagulant use; LS Mean Difference = -1.190, 95% CI 2-sided [-1.948 to -0.432] — LS Mean Difference is 5 mg daily minus weekly treatment

25. Secondary Outcome: Percent Change From Baseline in Greater Trochanter BMD, Week 104 / Endpoint
Time Frame: Week 104 / Endpoint
Population: ITT Population. Last Observation Carried Forward at Week 104.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent Change
Arm/Group | 5 mg Before Breakfast | 35 mg After Breakfast | 35 mg Before Breakfast
Number analyzed (Participants) | 279 | 274 | 280
Percent Change | 2.772 [2.255 to 3.289] | 3.691 [3.169 to 4.213] | 3.828 [3.312 to 4.344]
Statistical Analysis 1: Comparison: 5 mg Before Breakfast vs 35 mg After Breakfast; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; ANOVA; Fixed effects for treatment, pooled center and anticoagulant use; LS Mean Difference = -0.919, 95% CI 2-sided [-1.655 to -0.184] — LS Mean Difference is 5 mg daily minus weekly treatment
Statistical Analysis 2: Comparison: 5 mg Before Breakfast vs 35 mg Before Breakfast; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; ANOVA; Fixed effects for treatment, pooled center and anticoagulant use; LS Mean Difference = -1.056, 95% CI 2-sided [-1.787 to -0.326] — LS Mean Difference is 5 mg daily minus weekly treatment

26. Secondary Outcome: Percent Change From Baseline Urine Type-I Collagen N-telopeptide/ Creatinine (NTX/Cr), Week 13, ITT Population
Time Frame: Week 13
Population: ITT Population
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent Change
Arm/Group | 5 mg Before Breakfast | 35 mg After Breakfast | 35 mg Before Breakfast
Number analyzed (Participants) | 278 | 273 | 275
Percent Change | -42.595 [-45.869 to -39.320] | -46.366 [-49.673 to -43.059] | -45.420 [-48.714 to -42.126]
Statistical Analysis 1: Comparison: 5 mg Before Breakfast vs 35 mg After Breakfast; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; ANOVA; Fixed effects for treatment, pooled center and anticoagulant use; Least Squares Mean Difference = 3.771, 95% CI 2-sided [-0.885 to 8.427] — LS Mean Difference is 5 mg daily minus weekly treatment
Statistical Analysis 2: Comparison: 5 mg Before Breakfast vs 35 mg Before Breakfast; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; ANOVA; Fixed effects for treatment, pooled center and anticoagulant use; Least Squares Mean Difference = 2.826, 95% CI 2-sided [-1.819 to 7.471] — LS Mean Difference is 5 mg daily minus weekly treatment

27. Secondary Outcome: Percent Change From Baseline Urine Type-I Collagen N-telopeptide / Creatinine (NTX / Cr), Week 26, ITT Population
Time Frame: Week 26
Population: ITT Population
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent Change
Arm/Group | 5 mg Before Breakfast | 35 mg After Breakfast | 35 mg Before Breakfast
Number analyzed (Participants) | 271 | 265 | 272
Percent Change | -43.075 [-46.449 to -39.702] | -45.705 [-49.119 to -42.291] | -47.692 [-51.062 to -44.323]
Statistical Analysis 1: Comparison: 5 mg Before Breakfast vs 35 mg After Breakfast; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; ANOVA; Fixed effects for treatment, pooled center and anticoagulant use; Least Squares Mean Difference = 2.630, 95% CI 2-sided [-2.171 to 7.431] — LS Mean Difference is 5 mg daily minus weekly treatment
Statistical Analysis 2: Comparison: 35 mg Before Breakfast; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; ANOVA; Fixed effects for treatment, pooled center and anticoagulant use; Least Squares Mean Difference = 4.617, 95% CI 2-sided [-0.152 to 9.386] — LS Mean Difference is 5 mg daily minus weekly treatment

28. Secondary Outcome: Percent Change From Baseline Urine Type-I Collagen N-telopeptide / Creatinine (NTX / Cr), Week 52, ITT Population
Time Frame: Week 52
Population: ITT Population
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent Change
Arm/Group | 5 mg Before Breakfast | 35 mg After Breakfast | 35 mg Before Breakfast
Number analyzed (Participants) | 256 | 253 | 257
Percent Change | -42.223 [-45.710 to -38.735] | -47.263 [-50.771 to -43.754] | -46.863 [-50.345 to -43.380]
Statistical Analysis 1: Comparison: 5 mg Before Breakfast vs 35 mg After Breakfast; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; ANOVA; Fixed effects for treatment, pooled center and anticoagulant use; Least Squares Mean Difference = 5.040, 95% CI 2-sided [0.091 to 9.989] — LS Mean Difference is 5 mg daily minus weekly treatment
Statistical Analysis 2: Comparison: 5 mg Before Breakfast vs 35 mg Before Breakfast; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; ANOVA; Fixed effects for treatment, pooled center and anticoagulant use; Least Squares Mean Difference = 4.640, 95% CI 2-sided [-0.293 to 9.574] — LS Mean Difference is 5 mg daily minus weekly treatment

29. Secondary Outcome: Percent Change From Baseline Urine Type-I Collagen N-telopeptide / Creatinine (NTX / Cr), Week 52 / Endpoint, ITT Population
Time Frame: Week 52 / Endpoint
Population: ITT Population. Last Observation Carried Forward at Week 52.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent Change
Arm/Group | 5 mg Before Breakfast | 35 mg After Breakfast | 35 mg Before Breakfast
Number analyzed (Participants) | 279 | 274 | 278
Percent Change | -40.227 [-43.773 to -36.680] | -46.599 [-50.180 to -43.017] | -44.630 [-48.185 to -41.075]
Statistical Analysis 1: Comparison: 5 mg Before Breakfast vs 35 mg After Breakfast; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; ANOVA; Fixed effects for treatment, pooled center and anticoagulant use; Least Squares Mean Difference = 6.372, 95% CI 2-sided [1.329 to 11.414] — LS Mean Difference is 5 mg daily minus weekly treatment
Statistical Analysis 2: Comparison: 35 mg After Breakfast vs 35 mg Before Breakfast; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; ANOVA; Fixed effects for treatment, pooled center and anticoagulant use; Least Squares Mean Difference = 4.403, 95% CI 2-sided [-0.619 to 9.425] — LS Mean Difference is 5 mg daily minus weekly treatment

30. Secondary Outcome: Percent Change From Baseline Urine Type-I Collagen N-telopeptide / Creatinine (NTX / Cr), Week 104, ITT Population
Time Frame: Week 104
Population: ITT Population.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent Change
Arm/Group | 5 mg Before Breakfast | 35 mg After Breakfast | 35 mg Before Breakfast
Number analyzed (Participants) | 242 | 234 | 236
Percent Change | -49.188 [-53.061 to -45.314] | -53.927 [-57.870 to -49.983] | -53.186 [-57.111 to -49.261]
Statistical Analysis 1: Comparison: 5 mg Before Breakfast vs 35 mg After Breakfast; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; ANOVA; Fixed effects for treatment, pooled center and anticoagulant use; LS Mean Difference = 4.739, 95% CI 2-sided [-0.793 to 10.271] — LS Mean Difference is 5 mg daily minus weekly treatment
Statistical Analysis 2: Comparison: 5 mg Before Breakfast vs 35 mg Before Breakfast; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; ANOVA; Fixed effects for treatment, pooled center and anticoagulant use; LS Mean Difference = 3.999, 95% CI 2-sided [-1.518 to 9.515] — LS Mean Difference is 5 mg daily minus weekly treatment

31. Secondary Outcome: Percent Change From Baseline Urine Type-I Collagen N-telopeptide / Creatinine (NTX / Cr), Week 104 / Endpoint, ITT Population
Time Frame: Week 104 / Endpoint
Population: ITT Population. Last Observation Carried Forward at Week 104.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent Change
Arm/Group | 5 mg Before Breakfast | 35 mg After Breakfast | 35 mg Before Breakfast
Number analyzed (Participants) | 279 | 274 | 278
Percent Change | -46.261 [-50.137 to -42.386] | -51.079 [-54.993 to -47.165] | -49.454 [-53.338 to -45.569]
Statistical Analysis 1: Comparison: 5 mg Before Breakfast vs 35 mg After Breakfast; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; ANOVA; Fixed effects for treatment, pooled center and anticoagulant use; LS Mean Difference = 4.817, 95% CI 2-sided [-0.693 to 10.327] — LS Mean Difference is 5 mg daily minus weekly treatment
Statistical Analysis 2: Comparison: 5 mg Before Breakfast vs 35 mg Before Breakfast; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; ANOVA; Fixed effects for treatment, pooled centers and anticoagulant use; LS Mean Difference = 3.192, 95% CI 2-sided [-2.295 to 8.680] — LS Mean Difference is 5 mg daily minus weekly treatment

32. Secondary Outcome: Percent Change From Baseline Serum Type-I Collagen C-telopeptide (CTX), Week 13, ITT Population
Time Frame: Week 13
Population: ITT Population
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent Change
Arm/Group | 5 mg Before Breakfast | 35 mg After Breakfast | 35 mg Before Breakfast
Number analyzed (Participants) | 280 | 275 | 277
Percent Change | -42.331 [-45.643 to -39.019] | -46.781 [-50.127 to -43.436] | -46.054 [-49.386 to -42.723]
Statistical Analysis 1: Comparison: 5 mg Before Breakfast vs 35 mg After Breakfast; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; ANOVA; Fixed effects for treatment, pooled center and anticoagulant use; Least Squares Mean Difference = 4.450, 95% CI 2-sided [-0.260 to 9.160] — LS Mean Difference is 5 mg daily minus weekly treatment
Statistical Analysis 2: Comparison: 5 mg Before Breakfast vs 35 mg Before Breakfast; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; ANOVA; Fixed effects for treatment, pooled center and anticoagulant use; Least Squares Mean Difference = 3.723, 95% CI 2-sided [-0.975 to 8.421] — LS Mean Difference is 5 mg daily minus weekly treatment

33. Secondary Outcome: Percent Change From Baseline Serum Type-I Collagen C-telopeptide (CTX), Week 26, ITT Population
Time Frame: Week 26
Population: ITT Population.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent Change
Arm/Group | 5 mg Before Breakfast | 35 mg After Breakfast | 35 mg Before Breakfast
Number analyzed (Participants) | 274 | 265 | 273
Percent Change | -44.386 [-47.882 to -40.889] | -49.183 [-52.743 to -45.623] | -49.358 [-52.863 to -45.852]
Statistical Analysis 1: Comparison: 5 mg Before Breakfast vs 35 mg After Breakfast; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; ANOVA; Fixed effects for treatment, pooled center and anticoagulant use; Least Squares Mean Difference = 4.798, 95% CI 2-sided [-0.195 to 9.790] — LS Mean Difference is 5 mg daily minus weekly treatment
Statistical Analysis 2: Comparison: 5 mg Before Breakfast vs 35 mg Before Breakfast; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; ANOVA; Fixed effects for treatment, pooled center and anticoagulant use; Least Squares Mean Difference = 4.972, 95% CI 2-sided [0.020 to 9.924] — LS Mean Difference is 5 mg daily minus weekly treatment

34. Secondary Outcome: Percent Change From Baseline in Serum Type-I Collagen C-telopeptide (CTX), Week 52, ITT Population
Time Frame: Week 52
Population: ITT Population
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent Change
Arm/Group | 5 mg Before Breakfast | 35 mg After Breakfast | 35 mg Before Breakfast
Number analyzed (Participants) | 258 | 256 | 258
Percent Change | -44.410 [-48.140 to -40.680] | -49.185 [-52.931 to -45.440] | -50.048 [-53.780 to -46.316]
Statistical Analysis 1: Comparison: 5 mg Before Breakfast vs 35 mg After Breakfast; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; ANOVA; Fixed effects for treatment, pooled center and anticoagulant use; Least Squares Mean Difference = 4.775, 95% CI 2-sided [-0.514 to 10.065] — LS Mean Difference is 5 mg daily minus weekly treatment
Statistical Analysis 2: Comparison: 5 mg Before Breakfast vs 35 mg Before Breakfast; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; ANOVA; Fixed effects for treatment, pooled center and anticoagulant use; Least Squares Mean Difference = 5.638, 95% CI [0.356 to 10.920] — LS Mean Difference is 5 mg daily minus weekly treatment

35. Secondary Outcome: Percent Change From Baseline in Serum Type-I Collagen C-telopeptide (CTX), Week 52 / Endpoint, ITT Population
Time Frame: Week 52 / Endpoint
Population: ITT Population. Last Observation Carried Forward at Week 52.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent Change
Arm/Group | 5 mg Before Breakfast | 35 mg After Breakfast | 35 mg Before Breakfast
Number analyzed (Participants) | 281 | 275 | 279
Percent Change | -42.172 [-45.959 to -38.385] | -48.724 [-52.556 to -44.892] | -47.703 [-51.506 to -43.901]
Statistical Analysis 1: Comparison: 5 mg Before Breakfast vs 35 mg After Breakfast; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; ANOVA; Fixed effects for treatment, pooled center and anticoagulant use; Least Squares Mean Difference = 6.552, 95% CI 2-sided [1.162 to 11.942] — LS Mean Difference is 5 mg daily minus weekly treatment
Statistical Analysis 2: Comparison: 5 mg Before Breakfast vs 35 mg Before Breakfast; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; ANOVA; Fixed effects for treatment, pooled center and anticoagulant use; Least Squares Mean Difference = 5.531, 95% CI 2-sided [0.164 to 10.897] — LS Mean Difference is 5 mg daily minus weekly treatment

36. Secondary Outcome: Percent Change From Baseline in Serum Type-I Collagen C-telopeptide (CTX), Week 104, ITT Population
Time Frame: Week 104
Population: ITT Population.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent Change
Arm/Group | 5 mg Before Breakfast | 35 mg After Breakfast | 35 mg Before Breakfast
Number analyzed (Participants) | 245 | 235 | 238
Percent Change | -44.155 [-48.803 to -39.506] | -51.985 [-56.737 to -47.232] | -52.538 [-57.257 to -47.818]
Statistical Analysis 1: Comparison: 5 mg Before Breakfast vs 35 mg After Breakfast; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; ANOVA; Fixed effects for treatment, pooled center and anticoagulant use; LS Mean Difference = 7.830, 95% CI 2-sided [1.175 to 14.485] — LS Mean Difference is 5 mg daily minus weekly treatment
Statistical Analysis 2: Comparison: 5 mg Before Breakfast vs 35 mg Before Breakfast; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; ANOVA; Fixed effects for treatment, pooled centers and anticoagulant use; LS Mean Difference = 8.383, 95% CI 2-sided [1.757 to 15.010] — LS Mean Difference is 5 mg daily minus weekly treatment

37. Secondary Outcome: Percent Change From Baseline in Serum Type-I Collagen C-telopeptide (CTX), Week 104 / Endpoint, ITT Population
Time Frame: Week 104 / Endpoint
Population: ITT Population. Last Observation Carried Forward at Week 104.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent Change
Arm/Group | 5 mg Before Breakfast | 35 mg After Breakfast | 35 mg Before Breakfast
Number analyzed (Participants) | 281 | 275 | 279
Percent Change | -41.451 [-45.960 to -36.942] | -49.253 [-53.815 to -44.691] | -48.752 [-53.279 to -44.224]
Statistical Analysis 1: Comparison: 5 mg Before Breakfast vs 35 mg After Breakfast; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; ANOVA; Fixed effects for treatment, pooled center and anticoagulant use; LS Mean Difference = 7.802, 95% CI 2-sided [1.385 to 14.220] — LS Mean Difference is 5 mg daily minus weekly treatment
Statistical Analysis 2: Comparison: 5 mg Before Breakfast vs 35 mg Before Breakfast; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; ANOVA; Fixed effects for treatment, pooled center and anticoagulant use; LS Mean Difference = 7.301, 95% CI 2-sided [0.911 to 13.690] — LS Mean Difference is 5 mg daily minus weekly treatment

38. Secondary Outcome: Percent Change From Baseline in Serum Bone-specific Alkaline Phosphatase, Week 13, ITT Population
Time Frame: Week 13
Population: ITT Population.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent Change
Arm/Group | 5 mg Before Breakfast | 35 mg After Breakfast | 35 mg Before Breakfast
Number analyzed (Participants) | 280 | 275 | 277
Percent Change | -23.386 [-25.425 to -21.347] | -25.141 [-27.201 to -23.082] | -25.191 [-27.243 to -23.140]
Statistical Analysis 1: Comparison: 5 mg Before Breakfast vs 35 mg After Breakfast; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; ANOVA; Fixed effects for treatment, pooled center and anticoagulant use; Least Squares Mean Difference = 1.755, 95% CI 2-sided [-1.145 to 4.655] — LS Mean Difference is 5 mg daily minus weekly treatment
Statistical Analysis 2: Comparison: 5 mg Before Breakfast vs 35 mg Before Breakfast; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; ANOVA; Fixed effects for treatment, pooled center and anticoagulant use; Least Squares Mean Difference = 1.805, 95% CI 2-sided [-1.087 to 4.698] — LS Mean Difference is 5 mg daily minus weekly treatment

39. Secondary Outcome: Percent Change From Baseline in Serum Bone-specific Alkaline Phosphatase, Week 26, ITT Population
Time Frame: Week 26
Population: ITT Population.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent Change
Arm/Group | 5 mg Before Breakfast | 35 mg After Breakfast | 35 mg Before Breakfast
Number analyzed (Participants) | 274 | 265 | 273
Percent Change | -31.273 [-33.311 to -29.236] | -33.680 [-35.755 to -31.606] | -32.582 [-34.625 to -30.540]
Statistical Analysis 1: Comparison: 5 mg Before Breakfast vs 35 mg After Breakfast; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; ANOVA; Fixed effects for treatment, pooled center and anticoagulant use; Least Squares Mean Difference = 2.407, 95% CI 2-sided [-0.502 to 5.316] — LS Mean Difference is 5 mg daily minus weekly treatment
Statistical Analysis 2: Comparison: 5 mg Before Breakfast vs 35 mg Before Breakfast; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; ANOVA; Fixed effects for treatment, pooled center and anticoagulant use; Least Squares Mean Difference = 1.309, 95% CI 2-sided [-1.576 to 4.194] — LS Mean Difference is 5 mg daily minus weekly treatment

40. Secondary Outcome: Percent Change From Baseline in Serum Bone-specific Alkaline Phosphatase, Week 52, ITT Population
Time Frame: Week 52
Population: ITT Population.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent Change
Arm/Group | 5 mg Before Breakfast | 35 mg After Breakfast | 35 mg Before Breakfast
Number analyzed (Participants) | 258 | 256 | 258
Percent Change | -31.895 [-34.132 to -29.658] | -33.450 [-35.696 to -31.204] | -33.507 [-35.745 to -31.269]
Statistical Analysis 1: Comparison: 5 mg Before Breakfast vs 35 mg After Breakfast; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; ANOVA; Fixed effects for treatment, pooled center and anticoagulant use; Least Squares Mean Difference = 1.555, 95% CI 2-sided [-1.617 to 4.727] — LS Mean Difference is 5 mg daily minus weekly treatment
Statistical Analysis 2: Comparison: 5 mg Before Breakfast vs 35 mg Before Breakfast; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; ANOVA; Fixed effects for treatment, pooled center and anticoagulant use; Least Squares Mean Difference = 1.612, 95% CI 2-sided [-1.556 to 4.779] — LS Mean Difference is 5 mg daily minus weekly treatment

41. Secondary Outcome: Percent Change From Baseline in Serum Bone-specific Alkaline Phosphatase, Week 52 / Endpoint, ITT Population
Time Frame: Week 52 / Endpoint
Population: ITT Population. Last Observation Carried Forward at Week 52.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent Change
Arm/Group | 5 mg Before Breakfast | 35 mg After Breakfast | 35 mg Before Breakfast
Number analyzed (Participants) | 281 | 275 | 279
Percent Change | -31.367 [-33.536 to -29.199] | -32.802 [-34.996 to -30.607] | -32.829 [-35.007 to -30.652]
Statistical Analysis 1: Comparison: 5 mg Before Breakfast vs 35 mg After Breakfast; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; ANOVA; Fixed effects for treatment, pooled center and anticoagulant use; Least Squares Mean Difference = 1.434, 95% CI 2-sided [-1.652 to 4.521] — LS Mean Difference is 5 mg daily minus weekly treatment
Statistical Analysis 2: Comparison: 5 mg Before Breakfast vs 35 mg Before Breakfast; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; ANOVA; Fixed effect for treatment, pooled center and anticoagulant use; Least Squares Mean Difference = 1.462, 95% CI 2-sided [-1.611 to 4.535] — LS Mean Difference is 5 mg daily minus weekly treatment

42. Secondary Outcome: Percent Change From Baseline in Serum Bone-specific Alkaline Phosphatase, Week 104, ITT Population
Time Frame: Week 104
Population: ITT Population.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent Change
Arm/Group | 5 mg Before Breakfast | 35 mg After Breakfast | 35 mg Before Breakfast
Number analyzed (Participants) | 245 | 235 | 238
Percent Change | -33.394 [-35.969 to -30.819] | -36.143 [-38.776 to -33.510] | -36.810 [-39.424 to -34.195]
Statistical Analysis 1: Comparison: 5 mg Before Breakfast vs 35 mg After Breakfast; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; ANOVA; Fixed effects for treatment, pooled center and anticoagulant use; LS Mean Difference = 2.749, 95% CI 2-sided [-0.938 to 6.436] — LS Mean Difference is 5 mg daily minus weekly treatment
Statistical Analysis 2: Comparison: 5 mg Before Breakfast vs 35 mg Before Breakfast; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; ANOVA; Fixed effects for treatment, pooled center and anticoagulant use; LS Mean Difference = 3.416, 95% CI 2-sided [-0.255 to 7.087] — LS Mean Difference is 5 mg daily minus daily treatment

43. Secondary Outcome: Percent Change From Baseline in Serum Bone-specific Alkaline Phosphatase, Week 104 / Endpoint, ITT Population
Time Frame: Week 104 / Endpoint
Population: ITT Population. Last Observation Carried Forward at Week 104.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent Change
Arm/Group | 5 mg Before Breakfast | 35 mg After Breakfast | 35 mg Before Breakfast
Number analyzed (Participants) | 281 | 275 | 279
Percent Change | -32.572 [-35.042 to -30.103] | -34.769 [-37.268 to -32.271] | -34.824 [-37.303 to -32.344]
Statistical Analysis 1: Comparison: 5 mg Before Breakfast vs 35 mg After Breakfast; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; ANOVA; Fixed effects for treatment, pooled center and anticoagulant use; LS Mean Difference = 2.197, 95% CI 2-sided [-1.318 to 5.711] — LS Mean Difference is 5 mg daily minus weekly treatment
Statistical Analysis 2: Comparison: 5 mg Before Breakfast vs 35 mg Before Breakfast; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; ANOVA; Fixed effects for treatment, pooled center and anticoagulant use; LS Mean Difference = 2.251, 95% CI 2-sided [-1.248 to 5.751] — LS Mean Difference is 5 mg daily minus weekly treatment

44. Secondary Outcome: Number of Patients With at Least One New Fractured Vertebra, Week 52
Time Frame: Week 52
Population: ITT Population
Measure: Number; unit: Participants
Arm/Group | 5 mg Before Breakfast | 35 mg After Breakfast | 35 mg Before Breakfast
Number analyzed (Participants) | 257 | 257 | 257
Participants | 2 | 2 | 3
Statistical Analysis 1: Comparison: 5 mg Before Breakfast vs 35 mg After Breakfast; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p = 1.0000, Fisher Exact; Relative Risk = 1.00, 95% CI 2-sided [0.14 to 7.05]
Statistical Analysis 2: Comparison: 5 mg Before Breakfast vs 35 mg Before Breakfast; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p = 1.0000, Fisher Exact; Relative Risk = 1.50, 95% CI 2-sided [0.25 to 8.90]

45. Secondary Outcome: Number of Patients With at Least One New Fractured Vertebra, Week 52 / Endpoint, ITT Population
Time Frame: Week 52 / Endpoint
Population: ITT Population. Last Observation Carried Forward at Week 52.
Measure: Number; unit: Participants
Arm/Group | 5 mg Before Breakfast | 35 mg After Breakfast | 35 mg Before Breakfast
Number analyzed (Participants) | 270 | 261 | 271
Participants | 2 | 2 | 3
Statistical Analysis 1: Comparison: 5 mg Before Breakfast vs 35 mg After Breakfast; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p = 1.0000, Fisher Exact; Relative Risk = 1.03, 95% CI 2-sided [0.15 to 7.29]
Statistical Analysis 2: Comparison: 5 mg Before Breakfast vs 35 mg Before Breakfast; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p = 1.0000, Fisher Exact; Relative Risk = 1.49, 95% CI 2-sided [0.25 to 8.87]

46. Secondary Outcome: Number of Patients With at Least One New Fractured Vertebra, Week 104, ITT Population
Time Frame: Week 104
Population: ITT Population.
Measure: Number; unit: Participants
Arm/Group | 5 mg Before Breakfast | 35 mg After Breakfast | 35 mg Before Breakfast
Number analyzed (Participants) | 244 | 233 | 237
Participants | 5 | 2 | 4
Statistical Analysis 1: Comparison: 5 mg Before Breakfast vs 35 mg After Breakfast; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.4505, Fisher Exact; Relative Risk = 0.42, 95% CI 2-sided [0.08 to 2.14]
Statistical Analysis 2: Comparison: 5 mg Before Breakfast vs 35 mg Before Breakfast; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p = 1.0000, Fisher Exact; Relative Risk = 0.82, 95% CI 2-sided [0.22 to 3.03]

47. Secondary Outcome: Number of Patients With at Least One New Fractured Vertebra, Week 104 / Endpoint, ITT Population
Time Frame: Week 104 / Endpoint
Population: ITT Population. Last Observation Carried Forward at Week 104.
Measure: Number; unit: Participants
Arm/Group | 5 mg Before Breakfast | 35 mg After Breakfast | 35 mg Before Breakfast
Number analyzed (Participants) | 274 | 265 | 273
Participants | 5 | 2 | 6
Statistical Analysis 1: Comparison: 5 mg Before Breakfast vs 35 mg After Breakfast; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.4505, Fisher Exact; Relative Risk = 0.41, 95% CI 2-sided [0.08 to 2.11]
Statistical Analysis 2: Comparison: 5 mg Before Breakfast vs 35 mg Before Breakfast; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.7719, Fisher Exact; Relative Risk = 1.20, 95% CI 2-sided [0.37 to 3.90]

48. Secondary Outcome: Number of Patients With No New Fractured Vertebra, Week 52
Time Frame: Week 52
Population: ITT Population
Measure: Number; unit: Participants
Arm/Group | 5 mg Before Breakfast | 35 mg After Breakfast | 35 mg Before Breakfast
Number analyzed (Participants) | 257 | 257 | 257
Participants | 255 | 255 | 254
Statistical Analysis 1: Comparison: 5 mg Before Breakfast vs 35 mg After Breakfast; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p = 1.0000, Fisher Exact; Relative Risk = 1.00, 95% CI 2-sided [0.14 to 7.05]
Statistical Analysis 2: Comparison: 5 mg Before Breakfast vs 35 mg Before Breakfast; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p = 1.0000, Fisher Exact; Relative Risk = 1.50, 95% CI 2-sided [0.25 to 8.90]

49. Secondary Outcome: Number of Patients With No New Fractured Vertebra, Week 52 / Endpoint
Time Frame: Week 52 / Endpoint
Population: ITT Population. Last Observation Carried Forward at Week 52.
Measure: Number; unit: Participants
Arm/Group | 5 mg Before Breakfast | 35 mg After Breakfast | 35 mg Before Breakfast
Number analyzed (Participants) | 270 | 261 | 271
Participants | 268 | 259 | 268
Statistical Analysis 1: Comparison: 5 mg Before Breakfast vs 35 mg After Breakfast; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p = 1.0000, Fisher Exact; Relative Risk = 1.03, 95% CI 2-sided [0.15 to 7.29]
Statistical Analysis 2: Comparison: 5 mg Before Breakfast vs 35 mg Before Breakfast; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p = 1.0000, Fisher Exact; Relative Risk = 1.49, 95% CI 2-sided [0.25 to 8.87]

50. Secondary Outcome: Number of Patients With No New Fractured Vertebra, Week 104
Time Frame: Week 104
Population: ITT Population
Measure: Number; unit: Participants
Arm/Group | 5 mg Before Breakfast | 35 mg After Breakfast | 35 mg Before Breakfast
Number analyzed (Participants) | 244 | 233 | 237
Participants | 239 | 231 | 233
Statistical Analysis 1: Comparison: 5 mg Before Breakfast vs 35 mg After Breakfast; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.4505, Fisher Exact; Relative Risk = 0.42, 95% CI 2-sided [0.08 to 2.14]
Statistical Analysis 2: Comparison: 5 mg Before Breakfast vs 35 mg Before Breakfast; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p = 1.0000, Fisher Exact; Relative Risk = 0.82, 95% CI 2-sided [0.22 to 3.03]

51. Secondary Outcome: Number of Patients With No New Fractured Vertebra, Week 104 / Endpoint
Time Frame: Week 104 / Endpoint
Population: ITT Population. Last Observation Carried Forward at Week 104.
Measure: Number; unit: Participants
Arm/Group | 5 mg Before Breakfast | 35 mg After Breakfast | 35 mg Before Breakfast
Number analyzed (Participants) | 274 | 265 | 273
Participants | 269 | 263 | 267
Statistical Analysis 1: Comparison: 5 mg Before Breakfast vs 35 mg After Breakfast; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.4505, Fisher Exact; Relative Risk = 0.41, 95% CI 2-sided [0.08 to 2.11]
Statistical Analysis 2: Comparison: 5 mg Before Breakfast vs 35 mg Before Breakfast; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.7719, Fisher Exact; Relative Risk = 1.20, 95% CI 2-sided [0.37 to 3.90]

ADVERSE EVENTS:
Time Frame: Treatment-emergent Adverse Events (TEAEs) included all Adverse Events (AEs) from the date of first dose of study drug until the patient's Week 52 visit, or until the date the patient exited from the study for those who withdrew prior to the Week 52 visit.
Arm/Group | 5 mg Before Breakfast | 35 mg After Breakfast | 35 mg Before Breakfast
Serious Adverse Events (participants affected / at risk) | 31/307 | 32/307 | 32/308
Other Adverse Events (participants affected / at risk) | 243/307 | 250/307 | 264/308
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 5 mg Before Breakfast (N=307) | 35 mg After Breakfast (N=307) | 35 mg Before Breakfast (N=308)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Angina Pectoris (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Antidiuretic Hormone Abnormality (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0)
Anxiety Disorder due to General Medical Condition (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Aortic Valve Stenosis (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Atrial Fibrillation (Cardiac disorders) | 0 (0) | 1 (6) | 1 (1)
Atrial Flutter (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Bacterial Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Benign Breast Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Benign Neoplasm of Adrenal Gland (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Bladder Transitional Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Body Mass Index Decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Breast Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0)
Breast Dysplasia (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Cardiac Arrest (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Carotid Artery Stenosis (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0)
Cerebrovascular Accident (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Cholecystitis Acute (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Cholecystitis Chronic (Hepatobiliary disorders) | 0 (0) | 1 (1) | 1 (1)
Cholecystitis Infective (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 1 (1)
Chondrolysis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Coronary Artery Disease (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Cystocele (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Cystoscopy Abnormal (Investigations) | 1 (1) | 0 (0) | 0 (0)
Deafness Unilateral (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Deep Vein Thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Device Dislocation (General disorders) | 0 (0) | 0 (0) | 1 (1)
Diverticulitis (Infections and infestations) | 1 (1) | 1 (1) | 1 (1)
ECG Signs of Myocardial Ischaemia (Investigations) | 0 (0) | 1 (1) | 0 (0)
Emotional Disorder (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Exercise Tolerance Decreased (General disorders) | 0 (0) | 0 (0) | 1 (1)
Female Genital Tract Fistula (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Femoral Neck Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Femur Fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0)
Fibula Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Gastric Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Guillain-Barre Syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Herpes Zoster (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Hiatus Hernia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Humerous Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1)
Hyperparathyroidism (Endocrine disorders) | 3 (3) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Hypertensive Heart Disease (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Inguinal Hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Intestinal Obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Ischaemic Stroke (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Joint Instability (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Lung Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Macular Degeneration (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Major Depression (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Melaena (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Mengitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Mitral Valve Incompetence (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Myocardial Infarction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Oedematous Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 1 (1)
Ovarian Cyst (Reproductive system and breast disorders) | 1 (1) | 1 (1) | 0 (0)
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Pancreatic Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Pancreatitis Acute (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Parapsoriasis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Parkinson's Disease (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Pelvic Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Peritonitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pneumococcal sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 3 (4) | 0 (0)
Procedural Pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Pulmonary Microemboli (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pyelonephritis acute (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Radius Fracture (Injury, poisoning and procedural complications) | 1 (1) | 2 (2) | 1 (2)
Renal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Renal Failure Acute (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Sigmoiditis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Sinuitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Spinal Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Stress Urinary Incontinence (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Superventricular Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Therapeutic Agent Toxicity (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Thoracic Vertebral Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Thrombophlebitis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Tibia Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Upper Limb Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Urinary Bladder Polyp (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Urinary Tract Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Uterine Prolapse (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Vaginal Prolapse (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Varicose Vein (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Vasculitis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Vertigo Positional (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Wound Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 5 mg Before Breakfast (N=307) | 35 mg After Breakfast (N=307) | 35 mg Before Breakfast (N=308)
Abdominal Discomfort (Gastrointestinal disorders) | 1 (1) | 3 (3) | 6 (8)
Abdominal Distension (Gastrointestinal disorders) | 4 (4) | 3 (3) | 2 (2)
Abdominal Pain (Gastrointestinal disorders) | 10 (11) | 19 (21) | 20 (23)
Abdominal Pain Lower (Gastrointestinal disorders) | 4 (4) | 6 (6) | 5 (5)
Abdominal Pain Upper (Gastrointestinal disorders) | 8 (9) | 11 (15) | 26 (37)
Alopecia (Skin and subcutaneous tissue disorders) | 2 (2) | 5 (5) | 2 (2)
Anaemia (Blood and lymphatic system disorders) | 3 (3) | 8 (8) | 3 (3)
Anxiety (Psychiatric disorders) | 5 (5) | 1 (1) | 5 (5)
Arrhythmia (Cardiac disorders) | 4 (4) | 1 (1) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 33 (38) | 29 (39) | 27 (33)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 5 (5) | 3 (3)
Asthenia (General disorders) | 6 (6) | 5 (5) | 5 (5)
Asthma (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 1 (3) | 1 (1)
Back Pain (Musculoskeletal and connective tissue disorders) | 27 (31) | 29 (36) | 29 (31)
Blood Parathyroid Hormone Increased (Investigations) | 3 (3) | 2 (3) | 7 (8)
Blood Pressure Increased (Investigations) | 3 (3) | 4 (5) | 1 (1)
Bone Pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (3) | 6 (6)
Bronchitis (Infections and infestations) | 20 (26) | 17 (25) | 21 (24)
Cataract (Eye disorders) | 7 (7) | 4 (6) | 6 (7)
Chest Pain (General disorders) | 5 (5) | 1 (1) | 2 (2)
Cholethiasis (Hepatobiliary disorders) | 2 (2) | 3 (3) | 5 (5)
Colonic Polyp (Gastrointestinal disorders) | 2 (2) | 1 (1) | 4 (4)
Conjunctivitis (Eye disorders) | 4 (4) | 1 (1) | 1 (1)
Constipation (Gastrointestinal disorders) | 11 (13) | 17 (17) | 17 (17)
Contusion (Injury, poisoning and procedural complications) | 14 (15) | 11 (12) | 8 (12)
Cough (Respiratory, thoracic and mediastinal disorders) | 10 (11) | 9 (9) | 6 (6)
Cystitis (Infections and infestations) | 12 (13) | 9 (12) | 6 (6)
Dental Caries (Gastrointestinal disorders) | 4 (4) | 2 (2) | 5 (5)
Depression (Psychiatric disorders) | 5 (5) | 6 (6) | 7 (7)
Dermatitis Allergic (Skin and subcutaneous tissue disorders) | 4 (4) | 5 (6) | 7 (7)
Diarrhea (Gastrointestinal disorders) | 19 (25) | 30 (32) | 21 (24)
Diverticulitis (Infections and infestations) | 4 (4) | 2 (2) | 3 (4)
Diverticulum Intestinal (Gastrointestinal disorders) | 1 (1) | 4 (4) | 2 (2)
Dizziness (Nervous system disorders) | 10 (10) | 10 (10) | 11 (12)
Drug Intolerance (General disorders) | 2 (2) | 5 (5) | 6 (6)
Dry Mouth (Gastrointestinal disorders) | 3 (3) | 0 (0) | 4 (4)
Dyslipidaemia (Metabolism and nutrition disorders) | 4 (4) | 2 (2) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 16 (19) | 18 (24) | 12 (15)
Fall (Injury, poisoning and procedural complications) | 16 (18) | 18 (20) | 11 (11)
Fatigue (General disorders) | 4 (4) | 7 (8) | 1 (1)
Flatulence (Gastrointestinal disorders) | 5 (5) | 4 (4) | 5 (5)
Foot Fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 4 (4)
Gastritis (Gastrointestinal disorders) | 6 (6) | 3 (3) | 4 (4)
Gastroenteritis (Infections and infestations) | 7 (7) | 9 (9) | 10 (10)
Gastrointestinal Pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 4 (10)
Gastrointestinal Viral Infection (Infections and infestations) | 2 (2) | 4 (5) | 4 (5)
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 9 (9) | 3 (3) | 11 (12)
Gingivitis (Gastrointestinal disorders) | 2 (3) | 5 (6) | 3 (3)
Haematoma (Vascular disorders) | 0 (0) | 4 (4) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 4 (4) | 7 (7) | 4 (4)
Headache (Nervous system disorders) | 18 (18) | 9 (9) | 14 (14)
Herpes Zoster (Infections and infestations) | 3 (3) | 8 (8) | 3 (3)
Hiatus Hernia (Gastrointestinal disorders) | 4 (5) | 3 (3) | 10 (10)
Hot Flush (Vascular disorders) | 0 (0) | 4 (4) | 2 (2)
Hyperchlorhydria (Gastrointestinal disorders) | 5 (6) | 2 (2) | 5 (6)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 6 (6) | 13 (13) | 9 (9)
Hyperparathyroidism (Endocrine disorders) | 4 (4) | 0 (0) | 1 (1)
Hyperparathyroidism Secondary (Endocrine disorders) | 1 (1) | 2 (2) | 5 (6)
Hypersensitivity (Immune system disorders) | 3 (3) | 2 (2) | 4 (4)
Hypertension (Vascular disorders) | 20 (23) | 20 (20) | 21 (22)
Hypoparathyroidism (Endocrine disorders) | 5 (5) | 2 (2) | 4 (4)
Influenza (Infections and infestations) | 23 (28) | 27 (33) | 25 (29)
Influenza Like Illness (General disorders) | 3 (3) | 3 (3) | 5 (5)
Insomnia (Psychiatric disorders) | 3 (3) | 2 (2) | 4 (4)
Joint Sprain (Injury, poisoning and procedural complications) | 2 (2) | 3 (3) | 5 (5)
Memory Impairment (Nervous system disorders) | 3 (3) | 4 (4) | 0 (0)
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 9 (9) | 5 (5) | 12 (16)
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 13 (13) | 13 (14) | 11 (12)
Myalgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 4 (6) | 5 (5)
Nasopharyngitis (Infections and infestations) | 24 (29) | 32 (38) | 38 (48)
Nausea (Gastrointestinal disorders) | 15 (17) | 12 (15) | 14 (16)
Neck Pain (Musculoskeletal and connective tissue disorders) | 6 (6) | 5 (5) | 8 (8)
Nephrolithiasis (Renal and urinary disorders) | 2 (3) | 4 (4) | 4 (5)
Oedema Peripheral (General disorders) | 2 (2) | 6 (7) | 6 (6)
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 2 (2) | 3 (3)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 10 (10) | 8 (8) | 5 (5)
Pain (General disorders) | 0 (0) | 3 (3) | 4 (4)
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 13 (14) | 17 (18) | 14 (16)
Palpitations (Cardiac disorders) | 1 (1) | 4 (4) | 1 (1)
Paraesthesia (Nervous system disorders) | 3 (3) | 4 (5) | 0 (0)
Periodontitis (Gastrointestinal disorders) | 5 (5) | 3 (3) | 3 (5)
Pharyngitis (Infections and infestations) | 7 (7) | 11 (12) | 12 (16)
Pneumonia (Infections and infestations) | 1 (1) | 6 (7) | 5 (5)
Procedural Pain (Injury, poisoning and procedural complications) | 4 (5) | 2 (2) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2) | 4 (4) | 4 (5)
Pyrexia (General disorders) | 1 (1) | 1 (1) | 5 (10)
Radius Fracture (Injury, poisoning and procedural complications) | 2 (2) | 5 (5) | 6 (7)
Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 4 (4) | 5 (5)
Rhinitis (Infections and infestations) | 2 (2) | 5 (5) | 1 (1)
Sciatica (Nervous system disorders) | 7 (7) | 5 (6) | 2 (2)
Sinusitis (Infections and infestations) | 8 (8) | 4 (6) | 3 (3)
Sleep Disorder (Psychiatric disorders) | 1 (1) | 1 (1) | 4 (4)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 4 (4) | 1 (1)
Supraventricular Extrasystoles (Cardiac disorders) | 0 (0) | 4 (4) | 1 (1)
Tendonitis (Musculoskeletal and connective tissue disorders) | 6 (6) | 8 (8) | 3 (6)
Tooth Infection (Infections and infestations) | 4 (4) | 1 (1) | 4 (4)
Upper Respiratory Tract Infection (Infections and infestations) | 9 (9) | 13 (13) | 12 (17)
Urinary Tract Infection (Infections and infestations) | 20 (21) | 21 (27) | 22 (29)
Varicose Vein (Vascular disorders) | 2 (2) | 1 (1) | 4 (4)
Vertigo (Ear and labyrinth disorders) | 7 (10) | 7 (7) | 3 (3)
Viral Infection (Infections and infestations) | 2 (2) | 4 (4) | 3 (3)
Vomiting (Gastrointestinal disorders) | 10 (10) | 15 (18) | 8 (12)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The findings of the study may be published in a scientific journal or presented at a scientific meeting. Before submitting the results of the study for publication or presentation, the Investigator will allow the sponsor 30 days in which to review and comment on the manuscript.